CLINICAL TRIAL: NCT02685735
Title: Predicting, Understanding, and Speeding Recovery After Total Knee Arthroplasty
Brief Title: Predicting, Understanding and Speeding Recovery After TKA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of continued funding support
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00032506; 5P01GM113852 (NIH)
Record Dates: First submitted 2015-06-01; First posted 2016-02-19 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2023-05

CONDITIONS: Pain; Total Knee Replacement; Total Hip Replacement
MeSH Terms: conditions — Pain | interventions — Gabapentin; Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Active Comparator): Subjects will be randomized, stratifying for norepinephrine serotonin reuptake inhibitor (NSRI) use, to equal number to receive gabapentin or placebo pills. Drug treatment will begin 2 weeks prior to surgery and continue 3 weeks afterwards. Subjects randomized to gabapentin will receive 900 mg/day for the first week, 1800 mg/day for the next 3 weeks, and 900 mg/day for the last week.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Subjects will be randomized, stratifying for norepinephrine serotonin reuptake inhibitor (NSRI) use, to equal number to receive gabapentin or placebo pills. Drug treatment will begin 2 weeks prior to surgery and continue 3 weeks afterwards.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Drug treatment will begin 2 weeks prior to surgery and continue 3 weeks afterwards. Subjects randomized to gabapentin will receive 900 mg/day for the first week, 1800 mg/day for the next 3 weeks, and 900 mg/day for the last week.
  Other Names: neurontin
  Arms: Gabapentin
Drug: Placebo — Drug treatment will begin 2 weeks prior to surgery and continue 3 weeks afterwards. Subjects randomized to gabapentin will receive 900 mg/day for the first week, 1800 mg/day for the next 3 weeks, and 900 mg/day for the last week.
  Other Names: Inert ingredient
  Arms: Placebo

SUMMARY:
The objective of this research study is to better understand patterns of recovery after Total Knee Arthroplasty (TKA) amd Total Hip Replacement (THA). The study will evaluate how pain, activity and cognitive (i.e., thinking style) responses determine patterns of recovery, and the study will evaluate the efficacy of gabapentin versus placebo for improving recovery after surgery.

DETAILED DESCRIPTION:
The investigators propose a two-site, longitudinal, double-blind, randomized clinical intervention study to examine three specific aims:

Aim 1: Characterize the dynamic pain experience, activity, and cognitive response after TKA and determine patterns of recovery in these domains

Aim 2: Test whether gabapentin alters time course of recovery after TKA or THA in a manner dependent on its interaction with pre-drug pupil diameter and preferred style in the catastrophizing-optimism dimension

Aim 3: Test whether gabapentin increases pupil diameter in patients undergoing TKA or THA who are on high dose opioids preoperatively and to examine whether opioid use moderates the associations in Aim 1

Primary Hypothesis: Novel variance beyond established associations in recovery from pain following TKA or THA surgery is accounted for by the interaction between pupil diameter and Cognitive-Affective (C-A) state, and this interaction predicts efficacy of gabapentin to speed recovery.

Key secondary hypotheses: Disability, impulsivity, and attentional deficits recover after TKA or THA surgery follow a log of time pattern, and are predicted by C-A state and its interaction with pupil diameter. Gabapentin increases resting pupil diameter in patients scheduled for TKA who are receiving high doses of opioids.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective total knee or hip replacement
* American Society of Anesthesiologists physical status 1-3
* Participants must be able to read and write English

Exclusion Criteria:

* Inability to complete questionnaires
* Pregnancy
* Litigation or workers compensation related to joint surgery
* For 250 subjects in primary analysis - taking < 100 mg morphine equivalents/day. For 50 subjects to test gabapentin's effect on pupil diameter - taking >100 mg morphine equivalents/day
* history of Raynaud's disease of the feet
* suffering from a psychotic disorder or a recent psychiatric hospitalization
* history of eye surgery or topical eye medications that would render pupillometry unreliable or would directly affect pupil diameter.
* any disorder that would affect pupil responsivity or prevent accuracy of pupillometry such as movement disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from June 2, 2016 to August 2, 2021 at the Orthopeadic Clinics of Atrium Wake Forest Baptist and Davie County facilities and May 9, 2017 to July 21, 2020 at Cleveland Clinic facilities. Change in clinical practice resulted in inability to recruit subjects on high doses of opioid preoperatively, so recruitment of 50 subject in Aim 3 which was intended to separately examine interactions in this population did not occur.
Pre-assignment Details: Enrollment occurred greater or equal to 2 weeks prior to surgery. A total of 76 individuals were excluded prior to assignment to groups during the period prior to surgery because of cancellation of the planned surgery.
Groups:
- Gabapentin: Subjects will receive gabapentin, 900 mg/day for the first week, 1800 mg/day for the next 3 weeks, and 900 mg/day for the last week. Treatment will begin 2 weeks prior to surgery and continue 3 weeks afterwards.
- Placebo: Subjects will receive placebo pills and the number of pills will be the same as gabapentin in the active treatment arm. Treatment will begin 2 weeks prior to surgery and continue 3 weeks afterwards.
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 135 | 139
Completed (These subjects completed and provide data for the primary analysis. The total completed for secondary analyses is 89 in the gabapentin group and 93 in the placebo group. The reason for not completing was failure to complete questionnaires on at least one of the three occasions that these were performed.) | 117 | 123
Not Completed | 18 | 16
Not completed — Surgery Cancelled | 4 | 9
Not completed — Adverse Event | 10 | 3
Not completed — Preop testing found to be incomplete | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 117 | 123 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (7.8) | 60.7 (9.1) | 60.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 71 | 131
  Male | 57 | 52 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 116 | 121 | 237
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 98 | 107 | 205
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 117 | 123 | 240
Worst daily pain [Mean (Standard Deviation); unit: units on a scale] — From daily diaries completed for 2 weeks prior to surgery in which the participant rated each day the worst pain in the past 24 hours with 0=no pain and 10=worst pain imaginable
  units on a scale | 4.78 (2.77) | 4.71 (2.31) | 4.75 (2.54)
Resting pupil diameter [Mean (Standard Deviation); unit: mm] — Pupil diameter measured using infrared video recording at rest in a constant, low ambient light, low ambient noise room and in the absence of stimulation
  mm | 6.1 (1.9) | 5.9 (1.8) | 6.0 (1.8)
Optimism/acceptance of pain to catastrophizing cognitive style [Mean (Standard Deviation); unit: units on a scale] — A unidimensional scale that represents a broader spectrum of cognitive style that ranges from optimism/acceptance of pain to catastrophizing, derived from the Life Orientation Test-R (LOT-R) and catastrophizing to pain (CATS) questionnaires. Values of the derived scale are presented as theta, approximately equivalent to a z-score, with a range of -3 to 3 with negative numbers indicating optimism and positive numbers indicating catastrophizing.
  units on a scale | -0.12 (1.0) | 0.00 (1.08) | 0.00 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Adjusted Trajectory Model for Pain Between Gabapentin and Placebo--Intercept
Description: Daily pain intensity report for each subject was fitted using growth curve model with parameters of intercept (modeled initial pain) and slope of change in natural log of time, adjusted for prognostic predictors for gabapentin and placebo group separately. The daily pain intensity was the WORST pain (not the average pain) in the past 24 hr on a scale where 0 is no pain and 10 is worst imaginable pain.
  Values represent an intercept of modeled worst daily pain on the first day after hospital discharge across all participants, extracted from the mixed effect model. The intercept is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: The first day after hospital discharge up to 5 days post surgery
Population: The intention-to-treat population included all randomized patients who had at least one baseline pupil measurement, received at least one dose of study drug, and provided at least one pain score after the day of surgery.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 117 | 123
score on a scale | 7.57 [7.17 to 7.88] | 7.52 [7.16 to 7.88]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; The estimates were conducted using a linear mixed effects model contrasting differences in the gabapentin group versus placebo. In all cases, these differences are adjusted for prognostic variables including baseline pain, age, sex, pupil diameter, and catastophizing-optimism construct; Test type: Superiority — A likelihood-ratio test for change in pain was conducted for each outcome comparing a model with and without gabapentin treatment group. A statistically significant result is interpreted as evidence to support that the gabapentin treatment impacts some element of change after surgery (i.e, intercept or slope); p = 0.882, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05

2. Secondary Outcome: Wisconsin Card Sort Task
Description: This is a physical card sorting game which measures attention to shifts in implicit rules as the game progresses. Perseverative errors are the number of sequential errors when rules of the game shift and reflect dysfunction of attention. This score ranges from 0 to 64 with larger numbers reflecting more dysfunction of attention.
Time Frame: Preoperative, 2 months after surgery, 6 months after surgery
Population: The total completed for this secondary outcome is 113 in the gabapentin group and 116 in the placebo group. The reason for not completing was failure to complete questionnaires on at least one of the three occasions that these were performed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 113 | 116
score on a scale
  Preoperative | 4 [-8 to 20] | 2 [-10 to 24]
  2 months after surgery | 10 [-4 to 42] | 8 [-10 to 40]
  6 months after surgery | 18 [-4 to 45] | 18 [-2 to 41]

3. Secondary Outcome: Iowa Gambling Task
Description: This is a computer based card game which assesses risk taking and impulsivity in which a score of -100 to 100 is calculated. Lower numbers indicate greater impulsiivity
Time Frame: Preoperative, 2 months after surgery, 6 months after surgery
Population: The total completed for this secondary outcome is 111 in the gabapentin group and 115 in the placebo group. The reason for not completing was failure to complete the task on at least one of the three occasions that these were performed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 111 | 115
score on a scale
  Preoperative | 8 [5 to 14] | 7 [5 to 10]
  2 months after surgery | 6 [4 to 10] | 6 [4 to 10]
  6 months after surgery | 5 [4 to 8] | 5 [4 to 8]

4. Secondary Outcome: Tampa Scale of Kinesiophobia
Description: This 17-question scale assesses the degree of fear of pain from joint movement and is commonly used in orthopedic injury or surgery studies. The scale ranges from 17 to 68 with 17 indicating no fear of movement and 68 indicating severe fear.
Time Frame: Preoperative, 2 months after surgery, 6 months after surgery
Population: The total completed for secondary analyses is 113 in the gabapentin group and 117 in the placebo group. The reason for not completing was failure to complete questionnaires on at least one of the three occasions that these were performed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 113 | 117
score on a scale
  Preoperative | 37 [33 to 41] | 38 [35 to 41]
  2 months after surgery | 36 [33 to 39] | 37 [34 to 40]
  6 months after surgery | 37 [34 to 40] | 36 [34 to 40]

5. Other Pre Specified Outcome: Biomarkers of Stress
Description: Blood and cerebrospinal fluid will be obtained and frozen for subsequent assessment of hormones, neurochemicals, and other secreted compounds indicative of stress. Analysis will be in the future and dependent upon new literature for ideal biomarkers.
Time Frame: Preoperative
Population: Data were not collected
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Biomarkers of Noradrenergic Functioning
Description: Blood and cerebrospinal fluid will be obtained and frozen for subsequent assessment of compounds reflecting noradrenergic functioning. Analysis will be in the future and dependent upon new literature for ideal biomarkers.
Time Frame: Preoperative
Population: Data were not collected
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Comparison of Adjusted Trajectory Model for Pain Between Gabapentin and Placebo-- Slope
Description: Daily pain intensity report for each subject was fitted using growth curve model with parameters of intercept (modeled initial pain) and slope of change in natural log of time, adjusted for prognostic predictors for gabapentin and placebo group separately. The daily pain intensity was the WORST pain (not the average pain) in the past 24 hr on a scale where 0 is no pain and 10 is worst imaginable pain.
  Slope is defined as change in pain . Values represent the slope of modeled worst daily pain (0-10 scale as described above) divided by the natural log of time (days) across all participants, extracted from the mixed effect model. The slope is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: Postoperative Day 1 through Postoperative Day 60
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale/ln(day)
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 117 | 123
score on a scale/ln(day) | -0.110 [-0.113 to -0.107] | -0.114 [-0.117 to -0.111]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; The estimates were conducted using a linear mixed effects model contrasting differences in the gabapentin group versus placebo. In all cases, these differences are adjusted for prognostic variables including baseline pain, age, sex, pupil diameter, and catastrophizing-optimism construct; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.137, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05

8. Primary Outcome: Effect Pupil Diameter, Catastrophizing-optimism Construct, and Gabapentin on Model Fit of the Trajectory of Change in Worst Daily Pain After Surgery
Description: Daily pain intensity report for each subject was fitted using growth curve model, adjusted for pre-specified prognostic predictors . The daily pain intensity was the WORST pain (not the average pain) in the past 24 hr on a scale where 0 is no pain and 10 is worst imaginable pain.
  Deviance values were calculated from the model fit with just pre-specified prognostic predictors (Model 1) and the model fit with these predictors plus pupil diameter, catastrophizing-optimism construct, gabapentin treatment and their interaction. Deviance is a goodness-of-fit statistic for a statistical model; it is often used for statistical hypothesis testing. It is a generalization of the idea of using the sum of squares of residuals (SSR) in ordinary least squares to cases where model-fitting is achieved by maximum likelihood. Deviance ranges from 0 to infinity. The smaller the number the better the model fits the sample data.
  Model fits were compared using Chi-squared test.
Time Frame: Postoperative Day 1 through Postoperative Day 60
Population: The intention-to-treat population included all randomized patients who had at least one baseline pupil measurement, received at least one dose of study drug, and provided at least one pain score after the day of surgery. The primary analysis, as pre-specified in the statistical analysis plan and upon which sample size was determined, tested whether growth curve model for change in pain over 2 months was better fit when group, pupil diameter, and cognitive construct scores were added.
Measure: Number; unit: unitless
Groups:
- Adjusted Daily Worst Pain Trajectory Model (Model 1): Pain scores over time were fit to a ln(time) change model, including pre-defined prognostic covariates (age, sex, surgery site, and study site). This model considered each predictor and its interaction with the ln(time).
- Pain Trajectory Model Plus Pupil, Cognitive Style, and Study Drug Factors (Model 2): A full model that used all of the predictors from Model 1 with the addition of the catastrophizing-optimism cognitive construct (Cats-Opt), the baseline pupil diameter (Pupil), and randomized study drug group assignment (Group). As in Model 1, this model considered each predictor and its interaction with the ln(time). The two-way and three-way interactions among these variables were also specified alone and in conjunction with ln(time).
Arm/Group | Adjusted Daily Worst Pain Trajectory Model (Model 1) | Pain Trajectory Model Plus Pupil, Cognitive Style, and Study Drug Factors (Model 2)
Number analyzed (Participants) | 240 | 240
unitless | 43604 | 343523
Statistical Analysis 1: Comparison: Adjusted Daily Worst Pain Trajectory Model (Model 1) vs Pain Trajectory Model Plus Pupil, Cognitive Style, and Study Drug Factors (Model 2); The null hypothesis (H0) is that modeled trajectory of change in pain intensity report after total hip or total knee arthroplasty does not differ between oral gabapentin and placebo in a manner dependent on its interaction with preferred cognitive style and pre-surgery pupil resting diameter . The alternative hypothesis (H1) is that there is a difference between the two groups which is dependent on these interactions; Test type: Superiority; p < 0.0001, Chi-squared; 14 degrees of freedom; A likelihood ratio test was conducted to compare these two models, conditional on the difference in the degrees of freedom in both models. A statistically significant likelihood ratio test would be interpreted as evidence that the three mechanistic predictors (Catastrophising-Optimism construct, Study Group, resting Pupil diameter) impact some aspect of the change in pain that occurs after surgery. If a statistically significant effect is observed, the individual interaction parameters will be interpreted

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year per participant
Description: Adverse events related to known effects of gabapentin (sedation, dizziness, nausea) were assessed daily via the daily digital diaries beginning two weeks prior to surgery (the time study drug began) and continuing for 3 weeks after surgery, when study drug was discontinued. Adverse events during hospitalization were captured via the electronic medical health record. Other adverse events were captured daily via digital diaries until 2 months after surgery, then at 6- and 12- month phone calls.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/135 | 1/139
Serious Adverse Events (participants affected / at risk) | 1/135 | 0/139
Other Adverse Events (participants affected / at risk) | 17/135 | 2/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=135) | Placebo (N=139)
Death (Cardiac disorders) | 1 (1) | 0 (0) — The participant was found dead at home on the morning of surgery. Because of a history of several serious cardiac disorders, the presumptive cause of death was cardiac arrest
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=135) | Placebo (N=139)
Somnolence (Nervous system disorders) | 10 (10) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to 240 rather than 250 participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02685735/Prot_004.pdf
  • Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT02685735/SAP_003.pdf
  • Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT02685735/ICF_002.pdf